CLINICAL TRIAL: NCT07353177
Title: Effects of Hyperthermic Intraperitoneal Chemotherapy on Postoperative Bowel Motility and Complications: A Single-Center Retrospective Study
Brief Title: Effects of HIPEC on Postoperative Bowel Motility and Complications
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Hongpeng Jiang, attending doctor, Peking University People's Hospital
Other Study IDs: 2025PHB566-001
Record Dates: First submitted 2025-12-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: HIPEC; Gastro Intestinal Cancer; Adhesion Prevention; Bowel Functions
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with PM or stage T4b who underwent surgery were included: Patient selection criteria would include all the following: 1) Karnofsky performance status (KPS) score >50; 2) stage T4b (American Joint Committee on Cancer [AJCC] 8th edition stage) or peritoneal metastasis was confirmed during or after surgery; 3) life expectancy >3 months; 4) peripheral white blood cell count ≥3,500/mm3 and platelet count ≥80,000/mm3; and 5) acceptable liver, renal, cardiovascular, pulmonary, and coagulation function, and other major organ functions were able to endure a major operation. The exclusion criteria were defined as follows: 1) Performance of emergency surgery due to intestinal obstruction or perforation; 2) a history of inflammatory bowel disease (IBD); and 3) two or more independent surgical procedures on the gastrointestinal tract.
- Patients diagnosed with PM or stage T4b who underwent surgery combined with HIPEC: Patient selection criteria, as previously published [26], would include all the following: 1) Karnofsky performance status (KPS) score >50; 2) stage T4b (American Joint Committee on Cancer [AJCC] 8th edition stage) or peritoneal metastasis was confirmed during or after surgery; 3) life expectancy >3 months; 4) peripheral white blood cell count ≥3,500/mm3 and platelet count ≥80,000/mm3; and 5) acceptable liver, renal, cardiovascular, pulmonary, and coagulation function, and other major organ functions were able to endure a major operation. The exclusion criteria were defined as follows: 1) Performance of emergency surgery due to intestinal obstruction or perforation; 2) a history of inflammatory bowel disease (IBD); and 3) two or more independent surgical procedures on the gastrointestinal tract.
  Interventions: Other: Hyperthermic Intraperitoneal Chemotherapy (HIPEC)

INTERVENTIONS:
Other: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) — HIPEC was performed after gastrectomy or hemicolectomy, alimentary tract reconstruction and wound closure. Catheters, including the inflow and outflow tubes, were crossly placed into the abdominal cavity prior to primary abdominal closure. The temperature probes were placed on the inflow and outflow catheter tips. HIPEC was administered for 1 hour with an automatic HIPEC device (Thermochem НТ-1000 (ThermaSolutions, Inc., USA)). Perfusate used was Ringer's solution (5-6 L) mixed with cisplatin 50 mg/m2, 5-fluorouracil 500mg/m2 or raltitrexed 3 mg/m2, and warmed to an inflow temperature of 44 ℃.
  Groups: Patients diagnosed with PM or stage T4b who underwent surgery combined with HIPEC

SUMMARY:
This retrospective cohort study was conducted at our institution, involving patients with gastric cancer, appendiceal mucinous neoplasm, or colon cancer who underwent CRS with or without HIPEC between January 2017 and December 2023.

Patient selection criteria would include all the following: 1) Karnofsky performance status (KPS) score >50; 2) stage T4b (American Joint Committee on Cancer [AJCC] 8th edition stage) or peritoneal metastasis was confirmed during or after surgery; 3) life expectancy >3 months; 4) peripheral white blood cell count ≥3,500/mm3 and platelet count ≥80,000/mm3; and 5) acceptable liver, renal, cardiovascular, pulmonary, and coagulation function, and other major organ functions were able to endure a major operation. The exclusion criteria were defined as follows: 1) Performance of emergency surgery due to intestinal obstruction or perforation; 2) a history of inflammatory bowel disease (IBD); 3) two or more independent surgical procedures on the gastrointestinal tract; and 4) who received postoperative enema. Patients were divided into two groups based on the treatment strategy: (1) surgery alone (No-HIPEC group); (2) surgery combined with HIPEC (HIPEC group).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric, appendiceal, or colon malignant tumors of stage T4b or peritoneal metastases;
* Karnofsky performance status (KPS) score >50;
* Life expectancy >3 months;
* Peripheral white blood cell count ≥3,500/mm3 and platelet count ≥80,000/mm3;
* Acceptable liver, renal, cardiovascular, pulmonary, and coagulation function, and other major organ functions were able to endure a major operation.

Exclusion Criteria:

* Emergency surgery due to intestinal obstruction or perforation;
* A history of inflammatory bowel disease (IBD);
* Two or more independent surgical procedures on the gastrointestinal tract;
* Postoperative enema.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Involving patients with gastric cancer, appendiceal mucinous neoplasm, or colon cancer who underwent gastrectomy or hemicolectomy surgery with or without HIPEC between January 2017 and December 2023.
Sampling Method: Probability Sample
Enrollment: 193 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to first defecation after surgery | Perioperative
Length of postoperative stay | Perioperative

SECONDARY OUTCOMES:
Incidence of postoperative complications | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university people's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Result] 1. Montori G, Coccolini F, Ceresoli M, Catena F, Colaianni N, Poletti E, Ansaloni L: The treatment of peritoneal carcinomatosis in advanced gastric cancer: state of the art. Int J Surg Oncol 2014, 2014:912418. 2. Zani S, Papalezova K, Stinnett S, Tyler D, Hsu D, Blazer DG, 3rd: Modest advances in survival for patients with colorectal-associated peritoneal carcinomatosis in the era of modern chemotherapy. J Surg Oncol 2013, 107(4):307-311. 3. Zhang JF, Lv L, Zhao S, Zhou Q, Jiang CG: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Combined with Surgery: A 12-Year Meta-Analysis of this Promising Treatment Strategy for Advanced Gastric Cancer at Different Stages. Ann Surg Oncol 2022, 29(5):3170-3186. 4. Patel M, Arora A, Mukherjee D, Mukherjee S: Effect of hyperthermic intraperitoneal chemotherapy on survival and recurrence rates in advanced gastric cancer: a systematic review and meta-analysis. Int J Surg 2023, 109(8):2435-2450. 5. Verwaal VJ, van Ruth S, de Bree E, van Sloothen GW, van Tinteren H, Boot H, Zoetmulder FA: Randomized trial of cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy and palliative surgery in patients with peritoneal carcinomatosis of colorectal cancer. J Clin Oncol 2003, 21(20):3737-3743. 6. Verwaal VJ, Bruin S, Boot H, van Slooten G, van Tinteren H: 8-year follow-up of randomized trial: cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy in patients with peritoneal carcinomatosis of colorectal cancer. Ann Surg Oncol 2008, 15(9):2426-2432. 7. Yan TD, Deraco M, Baratti D, Kusamura S, Elias D, Glehen O, Gilly FN, Levine EA, Shen P, Mohamed F et al: Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy for malignant peritoneal mesothelioma: multi-institutional experience. J Clin Oncol 2009, 27(36):6237-6242.